CLINICAL TRIAL: NCT06360575
Title: MATCH Treatment Subprotocol C2: Crizotinib in Patients With Tumors With MET Exon 14 Deletion
Brief Title: Testing Crizotinib as Potentially Targeted Treatment in Cancers With MET Exon 14 Deletion Genetic Changes (MATCH - Subprotocol C2)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01127; NCI-2024-01127 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-C2 (Other: ECOG-ACRIN Cancer Research Group); EAY131-C2 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-04-10; First posted 2024-04-11 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — Biopsy; Specimen Handling; Crizotinib; X-Rays

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Crizotinib) (Experimental): Patients receive crizotinib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy on study and undergo radiologic evaluation and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Crizotinib; Procedure: Radiologic Examination

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Crizotinib — Given PO
  Other Names: Alkixen; Crizocent; MET Tyrosine Kinase Inhibitor PF-02341066; PF 02341066; PF-02341066; PF-2341066; PF02341066; Xalkori
Procedure: Radiologic Examination — Undergo radiologic evaluation
  Other Names: Radiologic Evaluation; Radiologic Exam

SUMMARY:
This phase II MATCH treatment trial tests how well crizotinib works to treat patients with cancers with MET exon 14 deletion genetic changes. Crizotinib is in a group of medications called tyrosine kinase inhibitors. It works by blocking enzymes that cancer cells need to grow and spread. It may also prevent the growth of new blood vessels that tumors need to grow.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive crizotinib orally (PO) twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy on study and undergo radiologic evaluation and blood sample collection throughout the study.

After completion of study treatment, patients followed up every 3 months for 2 years then every 6 months for year 3.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol EAY131/ NCI-2015-00054 prior to registration to treatment subprotocol
* Patient must fulfill all eligibility criteria outlined in Section 3.1 of MATCH Master protocol (excluding Section 3.1.6) at the time of registration to treatment step (Step 1, 3, 5, 7)
* Patient must have MET exon 14 skipping as defined via the MATCH Master Protocol and described or other mutations that disrupt exon 14 that are approved as a dynamic aMOI
* Patients must have an electrocardigram (ECG) within 8 weeks prior to treatment assignment and must not have clinically important abnormalities in rhythm, conduction or morphology of resting ECG, including complete left bundle branch block, third degree heart block
* Patients must not have known hypersensitivity to crizotinib or compounds of similar chemical or biologic composition
* Patient must not have had any of the following prior therapies: AMG 337, BMS 777607, cabozantinib (XL184), crizotinib (PF02341066), EMD1214063, foretinib (GSK1363089) (XL880), golvatinib (E7050), IncB28060 (INC280), JNJ 8877605, MGCD265, MK2461, MSC2156119J, PF 04217903, SGX523, tivantinib (ARQ197) or any other novel MET TKI with any MET inhibitory activity half-maximal inhibitory concentration (IC50) < 1 uM. Prior anti-HGF or anti-MET antibodies are acceptable
* Patients must not have a history of extensive disseminated/bilateral or known presence of grade 3 or 4 interstitial fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis, and pulmonary fibrosis, but not history of prior radiation pneumonitis
* Patients must not have had myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack within 3 months prior to start of study treatment. Clinically significant gastrointestinal (GI) abnormalities that may alter absorption (e.g., malabsorption syndrome, major resection of stomach or small bowel)
* Patients using drugs or foods that are known strong CYP3A4 inhibitors or inducers will be excluded. Patients must not require concurrent use of CYP3A substrates with narrow therapeutic indices
* Patients must not have had major surgery or tumor embolization within 4 weeks and minor surgery within 2 weeks prior to the initiation of the study drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-05-30 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. 90% two-sided confidence interval is calculated for ORR. For the purposes of this study, patients should be re-evaluated for response:
  * For treatments given in 21 day (3 week) cycles: every 3 cycles (9 weeks) for the first 33 cycles, and every 4 cycles thereafter (12 weeks)
  * For treatments given in 28 day (4 week) cycles: every 2 cycles (8 weeks) for the first 26 cycles, and every three cycles thereafter (12 weeks)
  * For treatments given in 42 day (6 week) cycles: every 2 cycles (12 weeks)

SECONDARY OUTCOMES:
Overall survival (OS) | From start of treatment that step until death, or censored at the date of last contact, assessed up to 3 years
  Will be evaluated specifically for each drug (or step). OS will be estimated using the Kaplan-Meier method.
6-month progression-free survival (PFS) rate | From start of treatment on that step until determination of disease progression or death from any cause, censored at the date of last disease assessment for patients who have not progressed, assessed at 6 months
  Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Progression free survival | From start of treatment on that step until determination of disease progression or death from any cause, censored at the date of last disease assessment for patients who have not progressed, assessed up to 3 years
  PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: David S Hong, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm